CLINICAL TRIAL: NCT06637384
Title: Effects of Hyaluronic Acid and Corticosteroid in Post Extraction Wound Healing of Diabetic Patients
Brief Title: Effect of Hyaluronic Acid and Single Dose Corticosteroid Injection to Improve Wound Healing in Controlled Diabetic Patients Post Tooth Extraction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rimsha Rasheed (Other)
Responsible Party: Sponsor-Investigator, Rimsha Rasheed, Dr. Rimsha Rasheed, University of Faisalabad
Organization: University of Faisalabad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Tuf/IRB/293/24
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus; Wound Healing Delayed
Keywords: Wound healing post extraction, Single dose corticosteroid, Diabetes Mellitus, Hyaluronic acid
MeSH Terms: conditions — Diabetes Mellitus | interventions — Hyaluronic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group 1 (No Intervention): The sockets untreated with hyaluronic acid and corticosteroid injection were designated as control group 1 where wound healing took place naturally via clot formation.
- Group 2 (Active Comparator): Patients treated with 0.2 % Hyaluronic acid (Gengigel Gingival Gel 20ml, Ricerfarma, Milan, Italy) applied in extraction socket.
  Interventions: Drug: Hyaluronic Acid (HA)
- Group 3 (Active Comparator): The extraction socket of these patients were treated with a single dose of Hy-Cortisone Injection 250 mg (Generic name: Hydrocortisone Sodium Succinate, Cirin Pharmaceuticals, Pakistan).
  Interventions: Drug: Corticosteroid Injection

INTERVENTIONS:
Drug: Hyaluronic Acid (HA) — Gengigel Gingival Gel 20ml, Ricerfarma, Milan, Italy
  Other Names: 0.2% Hyaluronic acid
  Arms: Group 2
Drug: Corticosteroid Injection — Hydrocortisone Sodium Succinate, Cirin Pharmaceuticals, Pakistan
  Arms: Group 3

SUMMARY:
The goal of this clinical trial is to learn if hyaluronic acid and corticosteroid improves wound healing in diabetic patients after oral extraction.

DETAILED DESCRIPTION:
After sample size estimation via Open Epi of 128, randomized clinical trial was performed on the patients from Oral and Maxillofacial Surgery Department in Madinah Teaching Hospital, Faisalabad. Patients were divided into three groups. Group 1 was subjected as control group, Group 2 was treated post extraction with 0.2 % Hyaluronic acid (Gengigel Gingival Gel 20ml, Ricerfarma, Milan, Italy) and Group 3 was treated with single dose Hy-Cortisone Injection 250 mg (Generic name: Hydrocortisone Sodium Succinate, Cirin Pharmaceuticals Pakistan) intramuscularly after extraction. Wound healing was assessed through Landry Healing Index. One-way ANOVA test was applied for comparative analysis and Post Hoc Tuckey's test was applied for pairwise comparisons between the groups

ELIGIBILITY:
Inclusion Criteria:

* • Controlled diabetic patients who had random blood glucose levels of 80 to 130 mg/dl, according to World Health Organization.

  * Age was defined from 25-55, irrespective of the gender.
  * Tooth extractions in maxilla or mandible without the presence of an acute infection or compromised periodontal state.

Exclusion Criteria:

* • Patients who declined to participate.

  * Patients below the age of 25 and above the age of 55.
  * Patients with uncontrolled diabetes mellitus (blood sugar levels high than the defined range)
  * Patients with history of adverse effects to local anesthetics or who are currently taking corticosteroids.
  * Patients with unmaintained oral hygiene and smoking habits.
  * Confirmation of any chronic illness, including those with hypertension or cardiac disorders.
  * Patients who have undergone any recent major surgical procedure.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Wound healing | 6 days
  The wound healing after follow was assessed via Landry Healing Index. This index had five grades very poor (1), poor (2), good (3), very good (4) and excellent (5). Each grade further had five parameters that included tissue color, response to palpation, granulation tissue, incision margin and suppuration.
  Tissue color was further categorized into >50% of red gingiva for grade 1 and 2. For grade 3 tissue color was specified as 25-50% of red gingiva. Less than 25% for grade 4 and all pink tissues for grade 5.Response to palpation was assessed as yes for grade 1 and 2, and no for the remaining three grades. The presence of granulation tissue was examined as yes for grade 1 and 2, and no for grade 3, 4 and 5. If the Incision margin was not epithelialized with loss of epithelium beyond incision margin it was considered grade 1. Incision margin not epithelialized with connective tissue exposure was marked as grade 2. For grade 3, 4 and 5, the connective tissue exposure was nil.

CONTACTS AND LOCATIONS:
Overall Officials: Rimsha Rasheed, BDS, MPhil Physiology, Principal Investigator — The University of Faisalabad
Locations (1):
- Department of Oral and Maxillofacial Surgery, Madinah Teaching Hospital, Faisalabad, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient data is kept confidential.

REFERENCES:
- See also: Implicates the role of hyaluronic acid in every major wound healing event. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7950635/
- See also: Describes the beneficial role of corticosteroid to reduce post operative pain and inflammation. — https://link.springer.com/article/10.1007/BF00542325